CLINICAL TRIAL: NCT05615532
Title: Effect of Injection Site on the Relative Bioavailability of Single Dose of LY3209590 and Evaluation of Absolute Bioavailability of LY3209590 in Healthy Participants
Brief Title: A Relative Bioavailability Study of LY3209590 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18222; I8H-MC-BDDD (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-11-10; First posted 2022-11-14 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Bioavailability; Injection sites

STUDY DESIGN:
Intervention Model Description: Part A is Parallel design and Part B is a crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- LY3209590 (Part A - Upper Arm) (Experimental): LY3209590 administered subcutaneously (SC) into the upper arm
  Interventions: Drug: LY3209590 (SC)
- LY3209590 (Part A - Thigh) (Experimental): LY3209590 administered SC into the thigh
  Interventions: Drug: LY3209590 (SC)
- LY3209590 (Part A - Abdominal Wall) (Experimental): LY3209590 administered SC into the abdominal wall
  Interventions: Drug: LY3209590 (SC)
- LY3209590 (Part B - IV Dose) (Experimental): LY3209590 administered intravenously (IV)
  Interventions: Drug: LY3209590 (IV)
- LY3209590 (Part B - SC Dose) (Experimental): LY3209590 administered SC into the abdominal wall
  Interventions: Drug: LY3209590 (SC)

INTERVENTIONS:
Drug: LY3209590 (SC) — Administered SC.
  Arms: LY3209590 (Part A - Abdominal Wall); LY3209590 (Part A - Thigh); LY3209590 (Part A - Upper Arm); LY3209590 (Part B - SC Dose)
Drug: LY3209590 (IV) — Administered IV.
  Arms: LY3209590 (Part B - IV Dose)

SUMMARY:
The study will be conducted in two parts (part A and part B). The main purpose of this study is to compare the amount of LY3209590 that gets into the blood stream and how long it takes the body to get rid of it, when self-administered at different body sites, abdominal wall, upper arm and thigh (part A), when administered by two different routes of injection, subcutaneously or intravenously (part B) in healthy participants.

The study may last up to 65 (part A) and 184 (part B) days, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who are overtly healthy as determined by medical evaluation
* Participants with body mass index (BMI) within the range 18.5 to 35.0 kilograms per meter squared (kg/m²)
* Male or female participants must agree to use contraception

Exclusion Criteria:

* Have a history of multiple or severe allergic reactions or a history of severe anaphylactic reaction
* Have known allergies to LY3209590, related compounds, or any components of the formulation
* Have an abnormality in the 12-lead electrocardiogram
* Intend to use prescription medication, including herbal medications and traditional medications
* Show evidence of human immunodeficiency virus infection or positive human immunodeficiency virus antibodies, hepatitis C or positive hepatitis C antibody, or hepatitis B or positive hepatitis B surface antigen
* Are lactating or pregnant

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Part A: Pharmacokinetics (PK): Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3209590 | Predose on Day 1 through Day 65
  Part A: PK: AUC0-∞ of LY3209590

SECONDARY OUTCOMES:
Part B: PK: AUC0-∞ of LY3209590 | Predose on Day 1 through Day 65
  Part B: PK: AUC0-∞ of LY3209590

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No